CLINICAL TRIAL: NCT02101619
Title: Assessment of Myocardial Tissue Damage in Aortic Stenosis for Risk Stratification
Brief Title: Assessment of Myocardial Tissue Damage in Aortic Stenosis
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Hari P. Chaliki M.D., MD, Mayo Clinic
Other Study IDs: 13-004385
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Aortic Stenosis
Keywords: aortic stenosis; myocardial tissue; echocardiography; MRI
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Moderate aortic stenosis.
- Severe aortic stenosis.

SUMMARY:
Aortic stenosis (AS) is the most common valve disease in the United States and most common indication for valve replacement surgery. Anatomical and hemodynamic severity of AS is insufficient for elucidating patients' prognosis. Therefore, the decision about the optimal timing of surgical intervention remains critical. However, the changes in structure and electrical activity of the cardiac muscle can be assessed by noninvasive imaging and electrocardiography (ECG). Degenerative myocardial changes characterized by fibrosis or collagen deposits are frequently observed in AS patients and have a negative impact on patient outcomes. In this project, our objective is to determine whether echocardiographic image analysis of integrated backscatter (IB), which can express changes in myocardial tissue composition (amount of fibrosis) based on its ultrasound reflectivity, global left ventricular (LV) load as measured by Zva, and ECG analysis of the duration of the QRS interval have a role in risk stratification for AS patients and to apply those methods to identify which patients would benefit from surgical intervention.

The investigators hypothesize that 1) the severity of myocardial damage can discriminate the prognosis in patients with AS, and 2) IB, Zva, and QRS interval can be diagnostic measures of the severity of myocardial damage. The investigators will measure the severity of myocardial fibrosis using MRI (reference) in 50 patients and will test the diagnostic significance of IB (testing method). Zva, QRS duration, and conventional echocardiographic measures will also be tested for diagnosing severity of myocardial fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe aortic stenosis determined by echocardiography
* Adults > 65 years old

Exclusion Criteria:

* Ejection fraction < 50%
* Valvular diseases of more than or equal to moderate degree other than aortic stenosis
* Prior myocardial infarction or coronary artery disease needs revascularization
* Atrial fibrillation (chronic)
* Pacemaker/defibrillator implanted
* Previous valve replacement performed
* Cardiomyopathy(HCM, infiltrative cardiomyopathy, constriction)
* Renal dysfunction (estimated GFR < 30ml/min/1.73m² or end stage renal failure)
* Patients with contraindication for MRI
* Patients with poor echocardiographic images

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients referred for echocardiography in Mayo Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2013-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Presence of myocardial fibrotic change determined by MRI. | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Hari Chaliki, MD, Principal Investigator — Mayo Clinic; Minako Katayama, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States